CLINICAL TRIAL: NCT06998446
Title: Sodium in the Skin and Atopic Dermatitis
Acronym: SIS-AD
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 22-38309; 1R01AR082831-01 (NIH)
Record Dates: First submitted 2025-05-12; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Eczema; Atopic Dermatitis
Keywords: Sodium; Salt
MeSH Terms: conditions — Eczema; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, microbiome skin swabs, and saliva will be collected during each in-person visit.
  After local anesthesia, one 6mm punch biopsy will be collected from patients with severe atopic dermatitis, from affected skin, for use in histopathology and/or cell culture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No History of AD: Healthy controls
- Mild AD: Eczema Area Severity Index (EASI): scores <7 will be considered mild AD
- Severe AD: Eczema Area Severity Index (EASI): scores >21 will be considered severe

SUMMARY:
The goal of this observational study is to understand factors associated with skin sodium storage in healthy adults and people with atopic dermatitis ages 50 and above.

The study is designed to test whether diet and skin barrier function are associated with skin sodium concentration and whether skin sodium concentration is linked to atopic dermatitis and immune profiles over time.

Participants will be asked to complete questionnaires, provide bio samples, and undergo non-contrast sodium MRI at 2-3 time points over 3-24 months.

DETAILED DESCRIPTION:
The central hypothesis of this proposal is that excess dietary sodium (consumed primarily as salt) is concentrated in the skin as a physiologic response to poor barrier function, and that high levels of skin sodium worsen atopic dermatitis.

The study will recruit 90 individuals (30 healthy participants, 30 with mild atopic dermatitis and 30 with severe atopic dermatitis) and follow them to identify factors associated with skin sodium storage. Diet will be evaluated using food frequency questionnaires and urine biomarkers, skin sodium concentration will be measured using a non-invasive sodium MRI technique, and atopic dermatitis activity and severity will be measured using multiple patient-reported outcomes and clinician scores. Participants without atopic dermatitis will be asked to visit the research site 4 times over 3 months. Participants with atopic dermatitis will be additionally asked to complete monthly severity scores for up to 24 months total and to visit the research site an additional 2 times when their disease severity changes.

The first specific aim will evaluate the association between dietary sodium intake and skin barrier function on skin sodium concentration. The primary analysis will use regression models to determine the association between dietary sodium intake and skin sodium concentration across 2-3 time points. The association with skin barrier function will also be evaluated.

The second specific aim will evaluate the extent to which skin sodium is associated with atopic dermatitis severity and persistence. The analysis will use regression models to determine the association between skin sodium and atopic dermatitis prevalence and severity. It will also examine immune profiles associated with skin sodium.

ELIGIBILITY:
Inclusion Criteria:

* Ages 50 years and above
* Willing to undergo non-contrast MRI (e.g., no contraindications to MRI, such as cardiac pacemakers, non-compatible intracranial vascular clips or pregnancy).

Exclusion Criteria:

* History of autoimmune disease.
* Cardiac events in the last six months.
* Impaired function of the liver or kidneys (glomerular filtration rate <60ml/min).
* Current use of medications that influence sodium excretion (e.g. thiazide diuretics, SGLT2 inhibitors and spironolactone), and/or chemotherapy or antibiotic treatment.
* Currently receiving phototherapy or taking systemic medications for atopic dermatitis including cyclosporine, methotrexate, or other broad immunosuppressive medications.

(Patients on dupilumab will not be excluded if they have been on dupilumab for at least two months and still meet the criteria for severe disease.)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Older adults with no history of atopic dermatitis, mild atopic dermatitis, or severe dermatitis.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Skin sodium concentration | 2 years
  Skin sodium concentration will be measured via non-contrast sodium MRI
Atopc dermatitis serverity | 2 years
  Atopic dermatitis severity will be measured via the eczema area severity index (EASI). The score range is 0-72 and higher scores indicate more severe atopic dermatitis.

SECONDARY OUTCOMES:
Atopic dermatitis severity and persistence | 2 years
  Atopic dermatitis severity and persistence will be tracked via assessments at clinic visits and via virtual monthly assessments using the Patient Oriented Eczema Measure (POEM). The POEM score ranges from 0-28 and higher scores indicate more severe atopic dematitis.
Atopic dermatitis severity | 2 years
  Atopic dermatitis-associated itch will be assessed at clinic visits using the numerical rating score for itch (NRS 11). The range for the NRS is 0-10, and higher scores indicate more severe itch / worse disease.
Atopic dermatitis severity | 2 years
  Atopic dermatitis severity will be measured at participant visits using the validated Investigator's Global Assessment (vIGA). The scores range from 0-4, and higher scores indicate more severe atopic dermatitis.
Atopic dermatitis severity | 2 years
  Atopic dermatitis severity will be measured at participant visits using a Body Surface Area (BSA) estimation. The BSA ranges from 0-100 and higher scores indicate more severe disease
Atopic dermatitis severity | 2 years
  Atopic dermatitis severity will be measured at participant visits using the Recap of Atopic Eczema (RECAP) measure of long term control. Scores range from 0-28, and higher scores indicate more severe atopic dermatitis.
Atopic dermatitis severity | 2 years
  Atopic dermatitis severity will be measured at participant visits using the Dermatology Life Quality Index (DLQI). Scores range from 0-30, and higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Katrina Abuabara, M.D., Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco VA Medical Center, San Francisco, California
  - UCSF Mt Zion Campus, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie the results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 1 year and ending 5 years after publication of the results
Access Criteria: Researchers interested in accessing data from the project must submit a written resource request via email to the Principal Investigator and sign a Data Use Agreement. De-identified data will be shared through a secure server.